CLINICAL TRIAL: NCT04548336
Title: Effects of Motor Imagery and Action Observation on Static and Dynamic Balance: A Randomized Controlled Trial
Brief Title: Mental Practice on Balance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Roy La Touche Arbizu, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: uammadrid33
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Movement, Involuntary
Keywords: Motor imagery
MeSH Terms: conditions — Dyskinesias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor Imagery (Experimental)
  Interventions: Behavioral: Motor Imagery
- Action Observation (Experimental)
  Interventions: Behavioral: Action observation
- Placebo group (Placebo Comparator)
  Interventions: Behavioral: Placebo group

INTERVENTIONS:
Behavioral: Motor Imagery — Motor imagery group will have to imagine motor gestures of static and dynamic balance
  Arms: Motor Imagery
Behavioral: Action observation — Action observation group will have to observe static and dynamic equilibrium motor gestures
  Arms: Action Observation
Behavioral: Placebo group — This group will watch a video of nature without a human component.
  Arms: Placebo group

SUMMARY:
The main objective of this research is to see the effect of two mental practice techniques on static and dynamic balance.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60
* Healthy and with no pain subjects

Exclusion Criteria:

* Any cognitive impairment that hindered viewing of audiovisual material.
* Difficulty understanding or communicating.
* Presence of systemic pathology, Central Nervous System or rheumatic disease.
* Inadequate understanding of the Spanish language to follow instructions for measuring and treatment.
* Collaboration of pregnant women.
* Underage subjects
* Subjects with pain at the time of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Posturography | Change in immediately at the end of the intervention.
  The device is a robotic device that evaluates motor function and consists of wirelessly sensed electromechanical platforms. This allows the evaluation of static and dynamic balance.

SECONDARY OUTCOMES:
Visual and Kinesthetic Motor Imagery Ability | Immediately before the intervention
  The degree of physical activity was objectified through the The International Physical Activity Questionnaire (IPAQ) questionnaire, which allows the subjects to be divided into three groups according to their level of activity, which can be high, moderate, and low or inactive. The IPAQ consists of 7 questions about the frequency, duration and intensity of activity (moderate and intense) performed in the last seven days, as well as walking and sitting time on a workday. The IPAQ scoring protocol assigns the following MET values to walking, moderate, and vigorous intensity activity: 3.3 METs, 4.0 METs, and 8.0 METs, respectively.
The degree of physical activity | Immediately before the intervention
  The degree of physical activity was objectified through the The International Physical Activity Questionnaire (IPAQ) questionnaire, which allows the subjects to be divided into three groups according to their level of activity, which can be high, moderate, and low or inactive. The IPAQ consists of 7 questions about the frequency, duration and intensity of activity (moderate and intense) performed in the last seven days, as well as walking and sitting time on a workday. The IPAQ scoring protocol assigns the following MET values to walking, moderate, and vigorous intensity activity: 3.3 METs, 4.0 METs, and 8.0 METs, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain